CLINICAL TRIAL: NCT03576794
Title: A Multicenter Randomized Placebo Controlled Treatment Study of Leflunomide in Polymyalgia Rheumatica
Brief Title: Treatment With Leflunomide in Patients With Polymyalgia Rheumatica
Acronym: PMRLEFRCT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elisabeth Brouwer (Other)
Collaborators: Dutch Arthritis Foundation Reuma Nederland (Unknown)
Responsible Party: Sponsor-Investigator, Elisabeth Brouwer, Principal investigator, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABR57022
Record Dates: First submitted 2018-04-17; First posted 2018-07-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Polymyalgia Rheumatica
Keywords: PMR RCT; Leflunomide
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Leflunomide; Prednisolone

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, placebo controlled treatment study during 12 months (part I) and an additional open-label follow-up of 12 months (part II).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leflunomide treatment (Active Comparator): Patients will receive prednisolone 15 mg once daily and will be randomized within 4 weeks of the start of glucocorticoid therapy (prednisolone). Prednisolon will be tapered according to a short fixed protocol with a slow gradual taper till 0 in week 27. During the first 2 weeks after randomization patients will receive Leflunomide 20 mg every other day in order to prevent early drug withdrawal due to side effects. After 2 weeks Leflunomide will be increased to 20 mg once daily and this therapy will be continued during 12 months.
  Interventions: Drug: Leflunomide 20 mg; Drug: Prednisolone
- Placebo control (Placebo Comparator): Patients will receive prednisolone 15 mg once daily and will be randomized within 4 weeks of the start of glucocorticoid therapy (prednisolone). Prednisolon will be tapered according to a short fixed protocol with a slow gradual taper till 0 in week 27. During the first 2 weeks after randomization patients will receive placebo 20 mg every other day in order to prevent early drug withdrawal due to side effects. After 2 weeks placebo will be increased to 20 mg once daily and this therapy will be continued during 12 months.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Leflunomide 20 mg — During the first 2 weeks after randomization patients will receive Leflunomide 20 mg every other day. After 2 weeks Leflunomide will be increased to 20 mg once daily and this therapy will be continued during 12 months.
  Arms: Leflunomide treatment
Drug: Prednisolone — Patients in both groups will receive prednisolone 15 mg once daily and will be randomized within 4 weeks of the start of glucocorticoid therapy (prednisolone). Prednisolon will be tapered according to a short fixed protocol with a slow gradual taper till 0 in week 27.

SUMMARY:
Over the last decades outcome has greatly improved for rheumatoid arthritis (RA) and spondyloarthritis (SpA). This is in sharp contrast to the situation for polymyalgia rheumatica (PMR), with a lifetime prevalence of 2.4% for women and 1.7% for men, PMR is the commonest auto-inﬂammatory musculoskeletal disease in adults aged ≥50 years. Due to population ageing, the number of PMR patients will likely double in the decades to come (CBS). Glucocorticoids (GC) are the mainstay of treatment. However, there is an unmet medical need of alternatives in the treatment of PMR as 50% of patients will relapse or have difficulties to reduce the corticosteroid doses. Also, there is increasing awareness of steroid related toxicity and in addition, long-term toxicity is a well-known side-effect of glucocorticoids in PMR.

Low dose methotrexate (< 10 mg per week) has been tested in two blinded randomized control trials and 4 open label studies and has shown low to moderate efficacy as corticosteroid-sparing agent. Studies on tumor necrosis factor (TNF) blockers yielded negative results. The effectiveness of leflunomide has only been convincingly demonstrated in case series.

The high rate of relapses and adverse events in steroid treated patients indicate that alternative adjuvant agents are needed.

There is evidence that leflunomide could serve as steroid sparing agent and that leflunomide can be used to prevent relapses in the clinical management of polymyalgia rheumatica.

We will perform a randomized placebo controlled trial. Eligible patients will be randomly assigned in a 1:1 ratio receiving either leflunomide 20 mg once daily + glucocorticoids , or placebo + glucocorticoids.

DETAILED DESCRIPTION:
Over the last decades outcome has greatly improved for rheumatoid arthritis (RA) and spondyloarthritis (SpA). This is in sharp contrast to the situation for polymyalgia rheumatica (PMR), with a lifetime prevalence of 2.4% for women and 1.7% for men, PMR is the commonest auto-inﬂammatory musculoskeletal disease in adults aged ≥50 years. Due to population ageing, the number of PMR patients will likely double in the decades to come (CBS). Glucocorticoids (GC) are the mainstay of treatment. However, there is an unmet medical need of alternatives in the treatment of PMR as 50% of patients will relapse or have difficulties to reduce the corticosteroid doses. Also, there is increasing awareness of steroid related toxicity and in addition, long-term toxicity is a well-known side-effect of glucocorticoids in PMR.

Low dose methotrexate (< 10 mg per week) has been tested in two blinded randomized control trials and 4 open label studies and has shown low to moderate efficacy as corticosteroid-sparing agent. Studies on TNF blockers yielded negative results. The effectiveness of leflunomide has only been convincingly demonstrated in case series.

The high rate of relapses and adverse events in steroid treated patients indicate that alternative adjuvant agents are needed.

There is evidence that leflunomide could serve as steroid sparing agent and that leflunomide can be used to prevent relapses in the clinical management of polymyalgia rheumatica.

We will perform a randomized placebo controlled trial. Eligible patients will be randomly assigned in a 1:1 ratio receiving either leflunomide 20 mg once daily + glucocorticoids , or placebo + glucocorticoids.

Primary endpoint The clinically relevant lower total number of relapses in leflunomide treated PMR patients as compared to placebo treated patients at 18 months.

Secondary endpoints

1. Steroid sparing capacity of leflunomide in patients with newly diagnosed PMR. Glucocorticoid sparing is expressed as a reduction of the cumulative glucocorticoid dose in the first 2 years of treatment.
2. Less time needed to reach both remission on glucocorticoids and glucocorticoid free remission
3. Less GC side effects in leflunomide PMR patient group

The first 2 weeks patients will receive leflunomide 20 mg every other day in order to prevent early drug withdrawal due to side effects. After 2 weeks leflunomide will be increased to 20 mg per day.

In case leflunomide has to be stopped due to side effects or inefficacy methotrexate will be used as rescue therapy 10 mg per week open label, based on the evidence that 10 mg methotrexate per week is steroid sparing. Those patients will be classified as non-responder.

Randomization will be stratified by age, gender and weight. Therefore, blocked randomization with variable block size will be performed.

Patients in both groups will be started on prednisolone 15 mg once daily and will be randomized within 2 weeks of the start of steroid therapy. The steroids will be tapered according to a short fixed protocol starting with 15 mg a day with a slow gradual taper till 0 in week 27.

Criteria for relapse or recurrence of PMR Relapse or recurrence will be measured according to an adaptation, based on expert opinion, to consensus criteria for PMR.

Relapse / recurrence Patient global higher than 3/ 10 and Physician global higher than 1/10 and An increased C reactive protein (CRP) ( > 5 mg/L) Is called a relapse if it was observed during steroid tapering, and is called a Recurrence if it was observed after steroid withdrawal.

Criteria for remission Patient global 3/ 10 or less and Physician global 1/10 or less and A normal CRP ( < 5 mg/L)

Secondary outcome measure PMR-AS The PMR-AS (Leeb and Bird) is a composite score with the following items: Physician global, Pt global, CRP, ability to raise the shoulders on examination, and duration of morning stiffness in minutes.

This randomized controlled trial (RCT) will assess:

1. Time to relapse and steroid-sparing capacity of leflunomide
2. PMR disease activity including patient reported outcome
3. Treatment related complications of steroids
4. Safety and tolerability of leflunomide

This blinded RCT in PMR is a unique study involving 5 centres in 4 different countries. It is the first study to use the recently developed consensus and outcome criteria in PMR which were developed by multidisciplinary groups including patients input. It is both timely and needed to fund a study in PMR since due to ageing in especially Western Europe the expectancy is that the incidence and prevalence of PMR will increase in the coming years. In brief: It is time to take PMR seriously and treat the patients with steroid sparing agents in order to prevent co-morbidities like diabetes, hypertension and osteoporosis in an ageing population.

The 5 centres (Department of Rheumatology and Immunology, Medical University Graz, Department of Rheumatology, Hospital of Southern Norway Trust Kristiansand, Kristiansand, Norway, The Department of Rheumatology, Southend University Hospital, Westcliff-on-sea, Chapel Allerton Hospital and St James's University Hospital Leeds and the University Medical Centre Groningen) participating in this study also set up an immediate early access outpatient clinic for PMR patients.

We will keep close contact with patients and their organizations to check whether our aims are in line with their expectations.

The relevance and gain for patients will be a different approach to PMR on the level of

* Early recognition/ making an appropriate diagnosis
* Starting steroid sparing treatment in an adequate dose at baseline
* Better outcome and earlier control of PMR with less relapses and cumulative dosis of steroids (benefit of thight control).

Our study can provide substantial benefit to the society. We seek to demonstrate that relatively cheap drug like leflunomide can improve the treatment of these PMR patients and limit the occurrence of relapses and GC-related side effects. Since leflunomide is an old and cheap drug the pharmaceutical companies are not interested in funding, we hope therefore that the Dutch Arthritis Association will fund our study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Female or male aged ≥ 50 years
3. PMR according to the American College of Rheumatology (ACR)/European league Against Rheumatism (EULAR) 2012 PMR core (essential) classification criteria
4. Newly diagnosed PMR being on glucocorticoids for less than 4 weeks

Exclusion Criteria:

1. Presence of any other connective tissue disease, including vasculitis/giant-cell arteritis
2. PMR on glucocorticoids for >4 week or >25 mg/day
3. History of alcohol or drug abuse or current alcohol or drug abuse
4. Transplanted organ (except corneal transplant performed more than 3 months prior to screening)
5. Evidence (as assessed by the investigator) of active infection, presence of hepatitis B surface antigen or hepatitis C antibody in blood, HIV positivity.
6. Malignancy within 5 years prior to screening, except for non-melanoma skin cancer
7. Exposure to DMARD/biological in the last 5 years
8. Pain syndromes, e.g. fibromyalgia, drug-induced myalgia
9. Active thyroid disease
10. Neurological diseases, e.g. Parkinson's disease
11. Contraindications for Leflunomide (serious immunodeficiency, e.g. AIDS, cytopenia as defined under 12, moderate to severe kidney failure (as defined under 12), liver test abnormality (as defined under 12)
12. Laboratory abnormalities:

    * Glomerular filtration rate <50 ml/min
    * Alanine-aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5x upper limit of normal
    * Platelet count <100 x 109/L (100,000/mm3)
    * Hemoglobin <85 g/L (8.5 g/dL; 5.3 mmol/L)
    * White blood cells <3.0 x 109/L (3,000/mm3)Absolute neutrophil count <2.0 x 109/L (2,000/mm3)
    * Absolute lymphocyte count <0.5 x 109/L (500/mm3)
13. Uncontrolled or poorly controlled hypertension
14. Major surgery or hospitalization within 3 month prior to screening
15. Any medical condition that could interfere with the implementation or interpretation of the study or with the safety of the patient during the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
PMR relapse | Within first 12 months of the study participation
  Relapse or recurrence will be measured according to an adaptation, based on expert opinion, to consensus criteria for PMR:
  * Patient global higher than 3/10 and
  * Physician global higher than 1/10 and
  * An increased CRP ( > 5 mg/L)
  It is called a "relapse" if it was observed during glucocorticoid tapering and is called a "recurrence" if it was observed after glucocorticoid withdrawal.

SECONDARY OUTCOMES:
Time till first relapse within first 24 months | Within first 24 months of the study participation
  Time measured in days
Percentage of patients with at least 1 relapse in the first 12 or 24 months | Within first 24 months of the study participation
  Percentage: patients with relapse in the first 12 or 24 months divided by total participating patients.
Number of relapsing patients within the first 24 months. | Within first 24 months of the study participation
Time till glucocorticoid free remission | Within first 24 months of the study participation
  Total days until patient has no glucocorticoid treatment and no signs of PMR.
Glucocorticoid-sparing effect | Within first 24 months of the study participation
  1. Glucocorticoid dose after 6, 12, 18 and 24 months.
  2. Cumulative glucocorticoid dose after 12, 18 and 24 months
Number of participants with adverse events and serious adverse events as assessed by MedDRA V21.0 | Within first 24 months of the study participation

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Brouwer, Principal Investigator — University Medical Center Groningen; E.M. Colin, Principal Investigator — ZGT Almelo
Locations (2):
- Netherlands (2):
  - ZGT Almelo, Almelo
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Yes
Manuscript after publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within 2 years after study termination, study data will be available and published
Access Criteria: Study data will be available upon request to the principal investigator

REFERENCES:
- [Background] Dasgupta B, Borg FA, Hassan N, Alexander L, Barraclough K, Bourke B, Fulcher J, Hollywood J, Hutchings A, James P, Kyle V, Nott J, Power M, Samanta A; BSR and BHPR Standards, Guidelines and Audit Working Group. BSR and BHPR guidelines for the management of giant cell arteritis. Rheumatology (Oxford). 2010 Aug;49(8):1594-7. doi: 10.1093/rheumatology/keq039a. Epub 2010 Apr 5. No abstract available. PMID 20371504
- [Background] Hernandez-Rodriguez J, Cid MC, Lopez-Soto A, Espigol-Frigole G, Bosch X. Treatment of polymyalgia rheumatica: a systematic review. Arch Intern Med. 2009 Nov 9;169(20):1839-50. doi: 10.1001/archinternmed.2009.352. PMID 19901135
- [Background] van der Veen MJ, Dinant HJ, van Booma-Frankfort C, van Albada-Kuipers GA, Bijlsma JW. Can methotrexate be used as a steroid sparing agent in the treatment of polymyalgia rheumatica and giant cell arteritis? Ann Rheum Dis. 1996 Apr;55(4):218-23. doi: 10.1136/ard.55.4.218. PMID 8733437
- [Background] Wagener P. [Methotrexate therapy of polymyalgia rheumatica]. Z Rheumatol. 1995 Nov-Dec;54(6):413-6. German. PMID 8578892
- [Background] Ferraccioli G, Salaffi F, De Vita S, Casatta L, Bartoli E. Methotrexate in polymyalgia rheumatica: preliminary results of an open, randomized study. J Rheumatol. 1996 Apr;23(4):624-8. PMID 8730115
- [Background] Feinberg HL, Sherman JD, Schrepferman CG, Dietzen CJ, Feinberg GD. The use of methotrexate in polymyalgia rheumatica. J Rheumatol. 1996 Sep;23(9):1550-2. PMID 8877923
- [Background] Caporali R, Cimmino MA, Ferraccioli G, Gerli R, Klersy C, Salvarani C, Montecucco C; Systemic Vasculitis Study Group of the Italian Society for Rheumatology. Prednisone plus methotrexate for polymyalgia rheumatica: a randomized, double-blind, placebo-controlled trial. Ann Intern Med. 2004 Oct 5;141(7):493-500. doi: 10.7326/0003-4819-141-7-200410050-00005. PMID 15466766
- [Background] Cimmino MA, Salvarani C, Macchioni P, Gerli R, Bartoloni Bocci E, Montecucco C, Caporali R; Systemic Vasculitis Study Group of the Italian Society for Rheumatology. Long-term follow-up of polymyalgia rheumatica patients treated with methotrexate and steroids. Clin Exp Rheumatol. 2008 May-Jun;26(3):395-400. PMID 18578959
- [Background] Catanoso MG, Macchioni P, Boiardi L, Pipitone N, Salvarani C. Treatment of refractory polymyalgia rheumatica with etanercept: an open pilot study. Arthritis Rheum. 2007 Dec 15;57(8):1514-9. doi: 10.1002/art.23095. PMID 18050171
- [Background] Salvarani C, Macchioni P, Manzini C, Paolazzi G, Trotta A, Manganelli P, Cimmino M, Gerli R, Catanoso MG, Boiardi L, Cantini F, Klersy C, Hunder GG. Infliximab plus prednisone or placebo plus prednisone for the initial treatment of polymyalgia rheumatica: a randomized trial. Ann Intern Med. 2007 May 1;146(9):631-9. doi: 10.7326/0003-4819-146-9-200705010-00005. PMID 17470831
- [Background] Kreiner F, Galbo H. Effect of etanercept in polymyalgia rheumatica: a randomized controlled trial. Arthritis Res Ther. 2010;12(5):R176. doi: 10.1186/ar3140. Epub 2010 Sep 20. PMID 20854662
- [Background] Lally L, Forbess L, Hatzis C, Spiera R. Brief Report: A Prospective Open-Label Phase IIa Trial of Tocilizumab in the Treatment of Polymyalgia Rheumatica. Arthritis Rheumatol. 2016 Oct;68(10):2550-4. doi: 10.1002/art.39740. PMID 27159185
- [Background] Devauchelle-Pensec V, Berthelot JM, Cornec D, Renaudineau Y, Marhadour T, Jousse-Joulin S, Querellou S, Garrigues F, De Bandt M, Gouillou M, Saraux A. Efficacy of first-line tocilizumab therapy in early polymyalgia rheumatica: a prospective longitudinal study. Ann Rheum Dis. 2016 Aug;75(8):1506-10. doi: 10.1136/annrheumdis-2015-208742. Epub 2016 Feb 29. PMID 26929219
- [Background] Adizie T, Christidis D, Dharmapaliah C, Borg F, Dasgupta B. Efficacy and tolerability of leflunomide in difficult-to-treat polymyalgia rheumatica and giant cell arteritis: a case series. Int J Clin Pract. 2012 Sep;66(9):906-9. doi: 10.1111/j.1742-1241.2012.02981.x. PMID 22897467
- [Background] Diamantopoulos AP, Hetland H, Myklebust G. Leflunomide as a corticosteroid-sparing agent in giant cell arteritis and polymyalgia rheumatica: a case series. Biomed Res Int. 2013;2013:120638. doi: 10.1155/2013/120638. Epub 2013 Sep 11. PMID 24106691
- [Background] Dasgupta B, Cimmino MA, Kremers HM, Schmidt WA, Schirmer M, Salvarani C, Bachta A, Dejaco C, Duftner C, Jensen HS, Duhaut P, Poor G, Kaposi NP, Mandl P, Balint PV, Schmidt Z, Iagnocco A, Nannini C, Cantini F, Macchioni P, Pipitone N, Del Amo M, Espigol-Frigole G, Cid MC, Martinez-Taboada VM, Nordborg E, Direskeneli H, Aydin SZ, Ahmed K, Hazleman B, Silverman B, Pease C, Wakefield RJ, Luqmani R, Abril A, Michet CJ, Marcus R, Gonter NJ, Maz M, Carter RE, Crowson CS, Matteson EL. 2012 Provisional classification criteria for polymyalgia rheumatica: a European League Against Rheumatism/American College of Rheumatology collaborative initiative. Arthritis Rheum. 2012 Apr;64(4):943-54. doi: 10.1002/art.34356. PMID 22389040
- [Background] Gran JT, Myklebust G. The incidence of polymyalgia rheumatica and temporal arteritis in the county of Aust Agder, south Norway: a prospective study 1987-94. J Rheumatol. 1997 Sep;24(9):1739-43. PMID 9292797
- [Background] Kermani TA, Warrington KJ. Polymyalgia rheumatica. Lancet. 2013 Jan 5;381(9860):63-72. doi: 10.1016/S0140-6736(12)60680-1. Epub 2012 Oct 8. Erratum In: Lancet. 2013 Jan 5;381(9860):28. PMID 23051717
- [Background] Matteson EL, Maradit-Kremers H, Cimmino MA, Schmidt WA, Schirmer M, Salvarani C, Bachta A, Dejaco C, Duftner C, Slott Jensen H, Poor G, Kaposi NP, Mandl P, Balint PV, Schmidt Z, Iagnocco A, Cantini F, Nannini C, Macchioni P, Pipitone N, Del Amo M, Espigol-Frigole G, Cid MC, Martinez-Taboada VM, Nordborg E, Direskeneli H, Aydin SZ, Ahmed K, Hazelman B, Pease C, Wakefield RJ, Luqmani R, Abril A, Marcus R, Gonter NJ, Maz M, Crowson CS, Dasgupta B. Patient-reported outcomes in polymyalgia rheumatica. J Rheumatol. 2012 Apr;39(4):795-803. doi: 10.3899/jrheum.110977. Epub 2012 Mar 15. PMID 22422492
- [Background] Dasgupta B, Borg FA, Hassan N, Barraclough K, Bourke B, Fulcher J, Hollywood J, Hutchings A, Kyle V, Nott J, Power M, Samanta A; BSR and BHPR Standards, Guidelines and Audit Working Group. BSR and BHPR guidelines for the management of polymyalgia rheumatica. Rheumatology (Oxford). 2010 Jan;49(1):186-90. doi: 10.1093/rheumatology/kep303a. Epub 2009 Nov 12. No abstract available. PMID 19910443
- [Background] Dejaco C, Singh YP, Perel P, Hutchings A, Camellino D, Mackie S, Abril A, Bachta A, Balint P, Barraclough K, Bianconi L, Buttgereit F, Carsons S, Ching D, Cid M, Cimmino M, Diamantopoulos A, Docken W, Duftner C, Fashanu B, Gilbert K, Hildreth P, Hollywood J, Jayne D, Lima M, Maharaj A, Mallen C, Martinez-Taboada V, Maz M, Merry S, Miller J, Mori S, Neill L, Nordborg E, Nott J, Padbury H, Pease C, Salvarani C, Schirmer M, Schmidt W, Spiera R, Tronnier D, Wagner A, Whitlock M, Matteson EL, Dasgupta B; European League Against Rheumatism; American College of Rheumatology. 2015 recommendations for the management of polymyalgia rheumatica: a European League Against Rheumatism/American College of Rheumatology collaborative initiative. Arthritis Rheumatol. 2015 Oct;67(10):2569-80. doi: 10.1002/art.39333. PMID 26352874
- [Background] Metzler C, Fink C, Lamprecht P, Gross WL, Reinhold-Keller E. Maintenance of remission with leflunomide in Wegener's granulomatosis. Rheumatology (Oxford). 2004 Mar;43(3):315-20. doi: 10.1093/rheumatology/keh009. Epub 2004 Jan 6. PMID 14963200